CLINICAL TRIAL: NCT05602363
Title: A Phase 1b Study of Oral AS-1763 in Patients With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma or Non-Hodgkin Lymphoma
Brief Title: AS-1763 in Patients With Previously Treated CLL/SLL or Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Carna Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C1763102
Record Dates: First submitted 2022-10-24; First posted 2022-11-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-07

CONDITIONS: B-cell Malignancy; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Waldenstrom Macroglobulinemia; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Follicular Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation (3+3 design) and determination of MTD and DLTs
  CLL/SLL or B-cell NHL patients will self-administer docirbrutinib oral tablet at multiple dose levels twice daily for 24 cycles (1 cycle = 28 days).
  Interventions: Drug: Docirbrutinib
- Dose Expansion (Experimental): Cohort 1: CLL/SLL patients, Cohort 2: B-cell NHL patients, Cohort 3: CLL/SLL or B-cell NHL patients with prior treatment with pirtobrutinib (Jaypirca) for an approved indication
  Patients will self-administer docirbrutinib oral tablet for 24 cycles (1 cycle = 28 days). Dose levels will be determined based on the result of dose escalation part.
  Interventions: Drug: Docirbrutinib

INTERVENTIONS:
Drug: Docirbrutinib — oral tablet, twice daily
  Other Names: AS-1763

SUMMARY:
This is an open-label, multi-center Phase 1b clinical study of oral AS-1763 (docirbrutinib) in patients with CLL/SLL or B-cell NHL who have failed or are intolerant to ≥2 lines of systemic therapy.

DETAILED DESCRIPTION:
This study consists of 2 parts.

Dose escalation part will enroll up to 27 patients to evaluate safety profile and tolerance of docirbrutinib using 3+3 design. The starting dose of docirbrutinib in oral tablet form is 100 mg twice daily (200 mg/day). Dose escalation will continue up to the planned maximum dose level or until the maximum tolerated dose (MTD) has been identified.

Dose expansion part will enroll up to 48 CLL/SLL patients (Cohort 1), up to 35 NHL patients (Cohort 2), and up to 10 patients with prior pirtobrutinib treatment for an approved indication (Cohort 3). The first 30 patients in each Cohort 1 or 2 will be allocated to three dose levels (n=10 at each dose level) which will be selected based on the data from dose escalation. Preliminary efficacy and safety data from the first 30 patients in one of cohorts will be used to identify the provisional recommended Phase 2 dose (RP2D) level. Thereafter, up to a further 18 patients for Cohort 1 and up to a further 5 patients for Cohort 2 will be enrolled and allocated to the provisional RP2D level. Cohort 3 will be enrolled in parallel with Cohorts 1 and 2 and will be allocated to up to two dose levels (either n=10 at a single dose level or n=5 at each of 2 dose levels).

Study assessments will continue for 24 cycles (1 cycle = 28 days) or until disease progression, occurrence of unacceptable toxicity, or discontinuation because of other reasons. Patients will then be followed for survival status for a further 2 years.

RP2D will be determined based on all the data generated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Provided written informed consent
* Histologically confirmed B-cell malignancy, including CLL/SLL, WM, MCL, MZL, or FL
* Patients with SLL, MCL, MZL, and FL: at least 1 radiographically measurable lesion
* Failed or are intolerant to ≥2 prior lines of systemic therapy
* ECOG Performance Status 0 to 2
* Adequate hematologic status (ie, absolute neutrophil count ≥0.75 × 10⁹/L, platelet count ≥50 × 10⁹/L, hemoglobin ≥8 g/dL) not requiring transfusion support or growth factors
* Adequate hepatic function
* Adequate renal function
* Ability to swallow tablets and comply with study requirements for the duration of study participation
* Male and female patients of reproductive potential: Willing to observe conventional and effective birth control methods
* Male patients: agree not to donate sperm during and for 6 months after the study
* Dose Expansion Cohort 3 patients: prior treatment with pirtobrutinib (Jaypirca) for an approved indication

Exclusion Criteria:

* Transformed disease (eg, Richter's transformation) prior to or during Screening
* Investigational agent or anticancer therapy within 5 half-lives before the planned start of docirbrutinib, except therapeutic monoclonal antibody treatment which must be discontinued at least 4 weeks before the start of docirbrutinib
* Current treatment with investigational therapy or planned investigational therapy which would be concurrent with this study
* Requiring therapeutic anticoagulation with warfarin
* Current treatment with certain strong CYP3A4 inhibitors or inducers
* Treatment with proton pump inhibitors within 7 days before first dose of docirbrutinib
* Current treatment with strong P-glycoprotein inhibitors or strong BCRP inhibitors
* Refractory to transfusion support
* Major surgery within 4 weeks before planned start of docirbrutinib
* Radiotherapy with a limited field of radiation for palliation within 7 days of the first dose of study treatment
* Any unresolved toxicities from prior therapy greater than NCI CTCAE Version 5.0 Grade 2 at the time of starting study treatment except for alopecia
* History of allogeneic or autologous stem cell transplant or CAR-T therapy within the last 30 days
* Active second malignancy unless in remission with life expectancy >2 years
* Known central nervous system (CNS) involvement by systemic lymphoma
* Active uncontrolled autoimmune cytopenia (eg, autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura) where new therapy introduced or concomitant therapy escalated within the 4 weeks before study enrollment is required to maintain adequate blood counts
* Clinically significant, uncontrolled cardiac, cardiovascular disease or history of myocardial infarction within 6 months before planned start of docirbrutinib, or prolongation of the QT interval corrected for heart rate using Fridericia's Formula (QTcF) >470 msec on at least 2 of 3 consecutive ECGs, and mean QTcF >470 msec on all 3 ECGs, during Screening
* Active uncontrolled systemic bacterial, viral, fungal, or parasitic infection
* Positive for HIV. For patients with unknown HIV status, HIV testing will be performed at Screening
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of docirbrutinib
* Pregnant or lactating.
* Known hypersensitivity to any component or excipient of docirbrutinib
* Prior treatment with docirbrutinib
* Dose Escalation and Cohort 3 patients: prior treatment with noncovalent BTKi except pirtobrutinib (Jaypirca)
* Dose Expansion Cohort 1 and Cohort 2 patients: prior treatment with any noncovalent BTKi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities (DLTs) and determination of maximum tolerated dose (MTD) | Up to 24 cycles (1 cycle = 28 days)
  Dose escalation
Overall response rate (ORR) as assessed by investigator | Up to 24 cycles (1 cycle = 28 days)
  Dose expansion

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) and clinical laboratory abnormalities | Up to 24 cycles (1 cycle = 28 days)
  Dose escalation, dose expansion
Area under the plasma concentration versus time curve (AUC) of docirbrutinib | Up to 24 cycles (1 cycle = 28 days)
  Dose escalation, dose expansion
Peak Plasma Concentration (Cmax) of docirbrutinib | Up to 24 cycles (1 cycle = 28 days)
  Dose escalation, dose expansion
Time to maximum plasma concentration (tmax) of docirbrutinib | Up to 24 cycles (1 cycle = 28 days)
  Dose escalation, dose expansion
ORR as assessed by investigator | Up to 24 cycles (1 cycle = 28 days)
  Dose escalation
Best overall response as assessed by investigator | Up to 24 cycles (1 cycle = 28 days)
  Dose expansion
Duration of response as assessed by investigator | Up to 24 cycles (1 cycle = 28 days)
  Dose expansion
Progression free survival as assessed by investigator | Up to 24 cycles (1 cycle = 28 days)
  Dose expansion
Overall survival | Up to 4 years
  Dose expansion

OTHER OUTCOMES:
Proportion of patients with BTK and PLCG2 gene mutation before and after disease progression | Up to 24 cycles (1 cycle = 28 days)
  Dose escalation, dose expansion

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - UC Irvine Health, Orange, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - American Oncology Partners, Fort Wayne, Indiana
  - University of Maryland Medical Center - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Optum Medical Care PC, Westbury, New York
  - Duke University, Durham, North Carolina
  - Taylor Cancer Research Center, Maumee, Ohio
  - Oncology Consultants, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No